CLINICAL TRIAL: NCT00607451
Title: A Double-blind, Placebo Controlled, Crossover, Ascending Single Dose Safety Tolerability, Pharmacokinetic and Pharmacodynamic Study of Neu-120 in Patients With Advanced Phase Idiopathic Parkinson's Disease With Levodopa Induced Dyskinesia
Brief Title: Safety, Tolerability, PK and PD Study of Neu-120 in the Treatment of Levodopa-induced Dyskinesia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Neurim Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PoC_12001; POC_120-CTIL
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Levodopa-induced Dyskinesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Neu-120
- 2 (Experimental)
  Interventions: Drug: Neu-120
- 3 (Experimental)
  Interventions: Drug: Neu-120
- 4 (Experimental)
  Interventions: Drug: Neu-120

INTERVENTIONS:
Drug: Neu-120 — Capsules of 300, 900 and 2700mg; administered as a single dose with a one week washout between each administration.

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetic and pharmacodynamic effects of single doses of Neu-120 in Parkinson's disease patients with levodopa-induced dyskinesia.

DETAILED DESCRIPTION:
Parkinson's disease is a progressive neurological disorder characterized by tremor, bradykinesia, rigidity, gait and postural instability and a variety of nonmotor symptoms. While levodopa effectively alleviates all symptoms of Parkinson's disease and restores motor function, within 3 to 5 years the majority of Parkinsonian patients develop levodopa-induced side effects, mainly dyskinesias (involuntary and uncontrolled movements such as twisting of a hand or a limb) and wearing off (progressive shortening of therapeutic response duration). Dyskinesias are the most disabling side effects of long term levodopa therapy in Parkinsonian patients. There is currently no approved drug for levodopa-induced dyskinesia.

The effects of three single ascending doses of orally administered Neu-120 will be evaluated in a double blind placebo controlled crossover proof of concept study. Following a 1-day screening visit, patients will be randomized to receive three single ascending doses of Neu-120 and placebo.

Patients will be admitted to the clinic on the evening prior to each visit on five occasions, each separated by 7 (-3) days. Levodopa challenges will be performed at baseline (visit 1) and at each treatment visit after withdrawal of all antiparkinsonian medications for 12 hours.

Blood samples will be taken for measurement of Neu-120 and levodopa plasma levels.

Primary parameter is improvement in levodopa-induced dyskinesia. Secondary parameters are safety, tolerability, pharmacodynamic assessments of dyskinesias and motor function, Neu-120/levodopa pharmacokinetic profiles and correlation between pharmacodynamic effects and Neu-120/levodopa levels.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 30-80 years old (both ages included).
* Use of adequate and effective birth control measures (not including the rhythm method) during the study period and up to 3 months after the end of study in men and women of child-bearing potential or within two years of menopause (these women will perform a urine pregnancy test at the screening visit)
* Idiopathic Parkinson Disease (UK PD Society Brain Bank Clinical Diagnosis Criteria) diagnosed for at least 3 years.
* Hoehn and Yahr "ON" time (good medication response) stage II-III.
* Treatment with levodopa at an optimized dose alone or with dopamine agonists, MAO-B inhibitors or COMT inhibitors that are stable for at least 4 weeks prior to visit 1
* Use of hypnotics, sedatives, beta-blockers, anxiolytics and antidepressant only if stable for at least 4 weeks prior to visit 1.
* A minimal baseline Levodopa induced dyskinesia score of 2 or more on question 32 (dyskinesias present during more than 25% of the waking day); a score of 2 or more on question 33 of UPDRS (severely disabling dyskinesias) Part IV (historical information).
* A minimal basal level of motor fluctuations of 25% or more cumulative hours of OFF time every day during waking hours on the UPDRS Part IV (a minimal score of 1 on question 39 of UPDRS, historical information).
* Patients have at least 33% motor improvement in response to their levodopa challenge dose based on UPDRS motor score (Part III) at visit 1.
* Patients experiencing peak-dose dyskinesia with a score of at least 2 on 2 or more (≥2) areas (a score of at least 4) on the modified AIMS scale in response to their levodopa challenge dose at visit 1.
* Patients must be in good general health as determined by medical history, physical examination, ECG, vital signs, serum biochemistry and haematology.
* Patients must have signed an informed consent form .

Exclusion Criteria:

* Patient has Non-idiopathic Parkinson's disease (e.g drug-induced or other form of secondary or atypical Parkinsonism).
* Neuropsychiatric exclusions: dementia (Mini Mental State Exam < 23, history or presence of psychosis (such as visual hallucinations while taking dopamine agonists), history of or current Axis I or Axis II mental disorders according to DSM-IV; severe depression (Hamilton scale > 17).
* Any clinically relevant acute or chronic diseases which could interfere with patients' safety during the trial, or expose them to undue risk, or which could interfere with the study objectives.
* History or presence of gastrointestinal, hepatic, or renal disease or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Pregnant or breast feeding women.
* Drug abuse or history of drug abuse (including alcohol), known drug addiction.
* Patients with severe postural hypotension (> 20 % variability between standing and supine).
* The following medications are forbidden for at least one month prior to visit 1 and during the course of the study: NMDA receptor antagonists (amantadine, memantine, budipine, dextromethorphan), medication with central dopaminergic antagonist activity (neuroleptics), CNS stimulants and sodium valproate (may exacerbate dyskinesias).
* Hoehn and Yahr score V when OFF (wheelchair-bound).
* The patient is participating in another study or has been participating in a study within the last 2 months.
* History of epilepsy and seizures.
* Any history of significant drug allergy.
* A history of unilateral or bilateral intracranial surgical procedures for Parkinson's Disease or any cerebral neurosurgery (except if occurred before the age of 18).
* History of severe pathology likely to recur during or immediately after the study.
* An inability to satisfactorily discontinue any study-forbidden medication.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-03; Primary Completion 2016-08-27 (Actual); Study Completion 2016-08-27 (Actual)

PRIMARY OUTCOMES:
Improving levodopa-induced dyskinesia | single day

SECONDARY OUTCOMES:
Safety and toleability | single dose

CONTACTS AND LOCATIONS:
Overall Officials: Tali Nir, Study Director — Neurim Pharmaceutical Ltd.
Locations (1):
- Neurim Pharmaceuticals Ltd., Tel Aviv, Israel